CLINICAL TRIAL: NCT00258544
Title: Microarray Analysis of Gene Expression in Idiopathic Pulmonary Fibrosis
Brief Title: Microarray Analysis of Gene Expression in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: MAA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kevin F. Gibson, Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY20070385
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Fibrosis
Keywords: Lung; Fibrosis; Idiopathic; Microarray; Tissue; Biopsy
MeSH Terms: conditions — Pulmonary Fibrosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Lung Tissue from a Lung Biopsy ordered by the patients physician. Also, a blood sample may be collected at the researchers discretion as listed in the addendum consent form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is investigating the way the lung is damaged in a condition called pulmonary fibrosis. Research studies will be conducted on lung tissue obtained from an open lung biopsy performed by the subject's surgeon. The identification of unique genetic markers of scarred lung may ultimately lead to new approaches to the diagnosis and treatment of pulmonary fibrosis.

DETAILED DESCRIPTION:
Subjects are being asked to participate in a research study that is investigating the way the lung is damaged in a condition called pulmonary fibrosis. These research studies are conducted in the laboratory on a portion of the tissue from the subject's lung biopsy that was performed by a surgeon. The lung biopsy is to be performed for clinical purposes to diagnose the cause of the subject's lung disease. The tissue used for the research study will in no way interfere with the ability of the pathologist to establish a diagnosis. In addition, the results of your breathing tests, chest X-rays and CT scans, and diagnosis made from the lung biopsy (and slides) will be collected. The goal of the study is to gain an understanding of the causes of pulmonary fibrosis and why it gets worse, which may ultimately lead to new therapies for this disease. Once the lung biopsies are obtained, the pathologist will examine the tissue and determine if there is a sufficient amount available to use in the study without compromising their ability to make a diagnosis. If so, the lung biopsy will be divided. One portion will be submitted to the research study and the other processed by the pathologist in the usual manner to make a diagnosis. The decision to use tissue for the research study will be at the complete discretion of the pathologists. The tissue used in the study will be further processed in the laboratory in order to analyze for the presence of genetic markers in the scarred tissue that are not present in normal. The identification of these unique genetic markers of scarred lung may ultimately lead to new approaches to the diagnosis and treatment of pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or age or older
* Diagnosis of pulmonary fibrosis
* Undergoing open lung biopsy

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population includes any patients seen at the Simmons Center for Interstitial Lung Disease with the possibility of having the diagnosis of Idiopathic Pulmonary Fibrosis who's physician has ordered an open Lung Biopsy. To check for the disease also known as IPF.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2001-10; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Microarray Analysis of Gene Expression in Idiopathic Pulmonary Fibrosis (IPF) | The time frame is open-ended with the goal of creating a bank of samples to support an indeterminant number of well phenotypes samples for studies of IPF.
  Microarray gene expression analysis involves the extraction of RNA from cells, synthesizing cDNA to hydridize to a probe array of genes, scanning signal intensities, and normalizing data to analyze probe-level expression for differential genes, Other methods of analyzing differential gene expression including Bulk RN-seq, and single cell RNA-seq will allow be employed where feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Gibson, MD, Principal Investigator — University of Pittsburgh - Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Pandit KV, Corcoran D, Yousef H, Yarlagadda M, Tzouvelekis A, Gibson KF, Konishi K, Yousem SA, Singh M, Handley D, Richards T, Selman M, Watkins SC, Pardo A, Ben-Yehudah A, Bouros D, Eickelberg O, Ray P, Benos PV, Kaminski N. Inhibition and role of let-7d in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2010 Jul 15;182(2):220-9. doi: 10.1164/rccm.200911-1698OC. Epub 2010 Apr 15. PMID 20395557
- See also: The Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease website. — http://www.upmc.com/Services/pulmonology/interstitial-lung-disease/Pages/default.aspx